CLINICAL TRIAL: NCT01534481
Title: Neurodevelopmental Effects of Donor Human Milk vs. Preterm Formula in Extremely Low Birth Weight (ELBW) Infants
Brief Title: Donor Milk vs. Formula in Extremely Low Birth Weight (ELBW) Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0047; U10HD021364 (NIH); U10HD040689 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027904 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD021373 (NIH); U10HD040492 (NIH); U10HD053109 (NIH); U10HD040461 (NIH); U10HD068244 (NIH); U10HD068263 (NIH); U10HD068278 (NIH); U10HD068284 (NIH); U10HD036790 (NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Infant, Newborn; Infant, Small for Gestational Age; Infant, Extremely Low Birth Weight
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Neurodevelopmental Impairment; Donor Breast Milk; Preterm Formula
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donor Milk (Active Comparator): Donor milk provided by the Human Milk Banking Association of North America
  Interventions: Biological: Donor Milk
- Preterm Formula (Placebo Comparator): Preterm formula determined by center practice
  Interventions: Dietary Supplement: Preterm Formula

INTERVENTIONS:
Biological: Donor Milk — Donor milk provided by the Human Milk Banking Association of North America
  Arms: Donor Milk
Dietary Supplement: Preterm Formula — Preterm Formula determined by center practice.
  Arms: Preterm Formula

SUMMARY:
The Milk Trial seeks to determine the effect on neurodevelopmental outcomes at age 22-26 months of donor human milk as compared to preterm infant formula as the in-hospital diet for infants whose mothers choose not to provide breast milk or are able to provide only a minimal amount. Infants will be randomized to receive donor breast milk or formula during their hospital stay. Infant's will be followed until they reach 22-26 months of age.

DETAILED DESCRIPTION:
There is strong evidence that maternal breast milk feedings in infancy confer multiple health benefits in the extremely preterm population (extremely low birth weight, ELBW, <1000 g). Studies suggest an IQ advantage of up to 8 points conferred by maternal milk feeding in this population. Rates of sepsis and necrotizing enterocolitis are also lower in human milk fed ELBW infants, and they experience shorter hospital stays and fewer re-hospitalizations in the first year of life. When mothers choose not to or are unable to provide milk, preterm formula is usually used. Recently, pasteurized donor human milk is available in some NICUs in the US as an alternative to preterm formula. Donor milk has not been well studied with regard to its safety and efficacy. It is unknown if donor human milk confers the same benefits as maternal milk with regard to neurodevelopmental and health outcomes. The proposed study will be the first US multicenter randomized trial of the health and developmental effects of donor milk as compared to preterm formula in ELBW infants receiving little or no maternal milk. Our long-term goal is to optimize neurodevelopmental and health outcomes for ELBW infants, maximizing their quality of life and societal functionality throughout their lives. If donor human milk has similar effects to maternal milk, the public health benefit of donor milk feedings in ELBW infants unable to receive maternal milk would be considerable.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 29 weeks.
* Admitted to the NICU at less than or equal to 72 hours of life
* Survived at least 12 hours

Exclusion Criteria:

* Chromosomal anomalies
* Cyanotic congenital heart disease
* Diagnosed intrauterine infection
* Other congenital disorders known to impair neurodevelopment
* NEC or IP prior to seeking consent
* Decision documented to limit intensive care therapies
* Congenital disorders that may affect feeding

Feeding Group Eligibility:

* Sole Diet Group: Infants will be eligible for the sole diet feeding protocol if the mother declines to provide breast milk for the baby.
* Supplemental Diet (minimal maternal milk) Group: Infants whose mothers initially choose to provide breast milk and begin pumping will be re-screened for eligibility at least weekly until the infant is 21 days old. If the mother stops expressing milk at any point prior to the infant's 21st day of life, her infant will be eligible for randomization. In addition, those whose mothers are providing less than 20% of the infant's dietary needs (averaged over past 5 days) when the infant reaches 21 days of age will be eligible for randomization at this point. No infant will be randomized after reaching 21 days.

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 483 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Colaizy, MD, MPH, Study Director — University of Iowa; Michele C Walsh, MD, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; C. Michael Cotten, MD, Principal Investigator — Duke University; David Carlton, MD, Principal Investigator — Emory University; Greg Sokol, MD, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P Van Meurs, MD, Principal Investigator — Stanford University; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Kristi L Watterberg, MD, Principal Investigator — University of New Mexico; Myra Wyckoff, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Jon Tyson, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Sara DeMauro, MD, Principal Investigator — University of Pennsylvania; Carl T D'Angio, MD, Principal Investigator — University of Rochester; Pablo J Sanchez, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov)

REFERENCES:
- [Derived] Colaizy TT, Poindexter BB, McDonald SA, Bell EF, Carlo WA, Carlson SJ, DeMauro SB, Kennedy KA, Nelin LD, Sanchez PJ, Vohr BR, Johnson KJ, Herron DE, Das A, Crawford MM, Walsh MC, Higgins RD, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network; MILK Trial Investigators; Ambalavanan N, Wyckoff MH, D'Angio CT, Bugg GW, Ohls RK, Reynolds AM, Sokol GM, Laptook AR, Olsen SL, White JR, Jadcherla SR, Bajaj M, Parimi PS, Schmidt B, Laughon MM, Barks J, Fisher KA, Hibbs AM, Peralta-Carcelen M, Cook N, Heyne RJ, Cavanaugh B, Adams-Chapman I, Fuller J, Hartley-McAndrew ME, Harmon HM, Duncan AF, Hines AC, Kilbride HW, Richards LA, Maitre NL, Natarajan G, Trembath AN, Carlson MD, Malcolm WF, Wilson-Costello DE; MILK Trial Investigators; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental Outcomes of Extremely Preterm Infants Fed Donor Milk or Preterm Infant Formula: A Randomized Clinical Trial. JAMA. 2024 Feb 20;331(7):582-591. doi: 10.1001/jama.2023.27693. PMID 38497706
- See also: NICHD NRN Website — https://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/overview.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Donor Milk: Pasteurized donor milk
- Formula: Preterm infant formula
Period: Overall Study
Arm/Group | Donor Milk | Formula
Started | 239 | 244
Complete Data for BSID III Cognitive Score at 22-26 Months | 175 | 192
Died After Discharge | 5 | 7
Died Before Discharge | 24 | 18
Survived to Discharge | 215 | 226
Completed (Death or BSID III cognitive score at 22-26 months) | 204 | 217
Not Completed | 35 | 27
Not completed — Lost to Follow-up | 29 | 24
Not completed — Incomplete Follow-up or No Study Data | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- DONORMILK: Pasteurized donor milk
- Total: Total of all reporting groups
Arm/Group | DONORMILK | FORMULA | Total
Number analyzed (Participants) | 239 | 244 | 483
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Age refers to the infant and is measured as gestational age in weeks
  weeks | 26 (1.8) | 26.1 (1.6) | 26 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 116 | 249
  Male | 106 | 128 | 234
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Black | 126 | 121 | 247
    Missing | 4 | 1 | 5
    Other | 11 | 14 | 25
    White | 98 | 108 | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 37 | 31 | 68
    Missing | 1 | 1 | 2
    Not Hispanic or Latino | 201 | 212 | 413
Weight of Infant at Birth [Mean (Standard Deviation); unit: grams] — Weight of the infant at birth, in grams
  grams | 848.6 (232) | 842.5 (219.8) | 845.5 (225.8)
Maternal Education [Count of Participants; unit: Participants] — Maternal education categories
  Participants
    College degree/more | 17 | 23 | 40
    High school degree | 82 | 93 | 175
    Less than high school degree | 64 | 57 | 121
    Missing | 19 | 17 | 36
    Partial college | 57 | 54 | 111

OUTCOME MEASURES:

1. Primary Outcome: Bayley Scales of Infant Development (BSID) Cognitive Composite Score
Description: Mean cognitive composite score (standardized mean 100, SD 15, range 54-145). Subjects who died prior to follow-up assigned the score of 54. (lower scores indicating greater impairment)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who died or were followed at 22-26 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 206 | 217
Score on a scale | 80.7 (17.4) | 81.1 (16.7)

2. Secondary Outcome: Total Deaths Before Discharge
Description: Infant died before discharge home.
Time Frame: From day of randomization to Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 1 year following birth
Population: The analysis population includes all randomized infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 239 | 244
Participants
  Death before discharge | 24 | 18
  Survival to discharge | 215 | 226

3. Secondary Outcome: Late Onset Sepsis (LOS)
Description: Number of infants diagnosed with LOS
Time Frame: From birth to Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 120 days following birth
Population: The analysis population includes all randomized infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 239 | 244
Participants
  Missing data | 1 | 0
  Late-onset sepsis | 47 | 37
  No late-onset sepsis | 191 | 207

4. Secondary Outcome: Necrotizing Enterocolitis (NEC)
Description: Number of infants diagnosed with NEC
Time Frame: as for outcome 3
Population: The analysis population includes all randomized infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 239 | 244
Participants
  Necrotizing enterocolitis | 10 | 22
  No necrotizing enterocolitis | 229 | 222

5. Secondary Outcome: Death or Necrotizing Enterocolitis (NEC)
Description: A composite outcome that measures the occurrence of death or NEC
Time Frame: as for outcome 3
Population: The analysis population includes all randomized infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 239 | 244
Participants
  Death or NEC | 27 | 33
  Survival without NEC | 212 | 211

6. Secondary Outcome: Change in Weight-for-age Z-score During Study
Description: Weight-for-age Z-scores were calculated at both baseline (study initiation) and study end (within one week of last study data collected) based on Fenton growth curves (2013). This outcome represents the change in weight-for-age Z-score during the course of the study (i.e., the Z-score at baseline was subtracted from the Z-score at study end).
  A value of 0 represents that the infant's weight-for-age Z-score is the same at the beginning and the end of the study. Positive values indicate the increase in the infant's weight-for-age Z-score during the study; negative values indicate the decrease in the infant's weight-for-age Z-score during the study.
Time Frame: During Study Intervention, the time between study randomization and discontinuation of study protocol. Infants exited from the study protocol 1-2 weeks prior to anticipated hospital discharge or 120 days, whichever is sooner
Population: The analysis population includes all randomized infants with non-missing data for weight at both the beginning and the end of the study.
Measure: Mean (Standard Deviation); unit: Change in Z-score (difference)
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 235 | 243
Change in Z-score (difference) | -0.4 (0.9) | -0.1 (0.9)

7. Secondary Outcome: Bayley Scales of Infant Development (BSID) Motor Composite Score
Description: Mean motor composite score (standardized mean 100, range 44-155). Subjects who died prior to follow-up assigned the score of 44. (lower scores indicating greater impairment)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who died or were followed at 22-26 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 202 | 213
Score on a scale | 80.3 (21.6) | 80.1 (19.9)

8. Secondary Outcome: Bayley Scales of Infant Development (BSID) Language Composite Score
Description: Mean language composite score (standardized mean 100, range 46-155). Subjects who died prior to follow-up assigned the score of 46. (lower scores indicating greater impairment)
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who died or were followed at 22-26 months.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 203 | 212
Score on a scale | 76.7 (19.6) | 75.8 (18.6)

9. Secondary Outcome: Moderate to Severe Cerebral Palsy
Description: Number of infants with moderate or severe grade of cerebral palsy
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who were followed (or adjudicated) at 22-26 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 188 | 199
Participants
  Missing data | 3 | 2
  Moderate-severe cerebral palsy | 14 | 20
  No moderate-severe cerebral palsy | 171 | 177

10. Secondary Outcome: Neurodevelopmental Impairment (NDI).
Description: Number of infants with NDI. NDI is defined as any of the following: Gross Motor Function Classification System score greater than or equal to 2, Bayley III cognitive or motor score less than 85 (1 standard deviation), Vision Impairment or Hearing impairment
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who were followed (or adjudicated) at 22-26 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 188 | 199
Participants
  Missing data | 11 | 10
  Neurodevelopmental impairment | 89 | 98
  No neurodevelopmental impairment | 88 | 91

11. Secondary Outcome: Profound Impairment
Description: Number of infants with profound impairment.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who were followed (or adjudicated) at 22-26 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 188 | 199
Participants
  Missing data | 4 | 5
  No profound NDI | 154 | 152
  Profound NDI | 30 | 42

12. Secondary Outcome: Death or Neurodevelopmental Impairment (NDI)
Description: A composite outcome that measures the occurrence of death through 22-26 months or NDI.
Time Frame: At 22-26 months corrected age
Population: The analysis population includes all randomized infants who died or were followed (or adjudicated) at 22-26 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Donor Milk | Formula
Number analyzed (Participants) | 217 | 224
Participants
  Missing data | 11 | 10
  Death or NDI | 118 | 123
  Survival without NDI | 88 | 91

ADVERSE EVENTS:
Time Frame: From day of randomization to Neonatal Research Network NRN infant status i.e., the first occurring of: discharge home, death, transfer, or 1 year following birth. For All-Cause Mortality, the time frame extends to follow-up (22-26 months) since deaths after discharge are included.
Arm/Group | Donor Milk | Formula
All-Cause Mortality (participants affected / at risk) | 29/239 | 25/244
Serious Adverse Events (participants affected / at risk) | 48/239 | 47/244
Other Adverse Events (participants affected / at risk) | 19/239 | 17/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Milk (N=239) | Formula (N=244)
Bradycardia neonatal (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Renal hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea neonatal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 13 (13) | 20 (21)
Neonatal intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neonatal intestinal perforation (Gastrointestinal disorders) | 4 (4) | 1 (5)
Pneumoperitoneum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neonatal cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
CNS ventriculitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 2 (2)
Disseminated aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 1 (1) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 14 (18) | 14 (14)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 2 (2)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neonatal hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 1 (1) | 0 (0)
Neonatal seizure (Nervous system disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure neonatal (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Labile blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Neonatal hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donor Milk (N=239) | Formula (N=244)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 2 (2) | 9 (9)
Acute on chronic liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Neonatal cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Neonatal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis neonatal (Infections and infestations) | 13 (15) | 6 (6)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neonatal hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 1 (1)
Neonatal seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Neonatal anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnea Neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension neonatal (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication Policies

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT01534481/Prot_SAP_000.pdf